CLINICAL TRIAL: NCT06535750
Title: Comparison Of The Effects Of Conventional Physiotherapy And Strengthening Exercises Additional To Conventional Physiotherapy On Pain, Muscle Strength, Joint Range Of Motion, Functionality And Quality Of Life In Patients With Rotator Cuff Syndrome
Brief Title: Comparison Of The Effects Of Conventional Physiotherapy And Strengthening Exercises With Rotator Cuff Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, assistant profesor, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBeykent-6
Record Dates: First submitted 2024-07-23; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Rotator Cuff Syndrome; Physiotherapy
Keywords: Rotator Cuff; Exercise; Pain
MeSH Terms: conditions — Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotator Cuff Patients with used to conventional rehabilitation (Experimental): Patients in the experimental group received strengthening exercises with theraband in addition to the standard treatment programme. This programme included the following:
  Strengthening Exercises: Low-row, biceps strengthening, shoulder horizontal abduction and shoulder horizontal adduction, external rotation. After the pain decreased, strengthening exercises for subscapularis, infraspinatus, supraspinatus, teres minor, deltoid and scapulothoracic muscles were performed. The colour of the Theraband was chosen between yellow, red, green, blue and red to the extent tolerated by the patient.
  Interventions: Other: Exercise
- Rotator Cuff Patients with used to conventional rehabilitation add to strenght exercise. (Experimental): Patients in the experimental group received strengthening exercises with theraband in addition to the standard treatment programme. This programme included the following:
  Strengthening Exercises: Low-row, biceps strengthening, shoulder horizontal abduction and shoulder horizontal adduction, external rotation. After the pain decreased, strengthening exercises for subscapularis, infraspinatus, supraspinatus, teres minor, deltoid and scapulothoracic muscles were performed. The colour of the Theraband was chosen between yellow, red, green, blue and red to the extent tolerated by the patient.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants were randomly divided into two treatment groups. There are 10 patients in each group. The patients in the control group received a standard treatment programme, while the patients in the experimental group received strengthening exercises with theraband in addition to the standard treatment programme. Treatment sessions for both groups lasted 50-55 minutes and were performed three days a week. Details of the study groups are given below.

SUMMARY:
Various options are available for the treatment of rotator cuff syndrome, including conservative and surgical. Conservative treatment methods include activity modification, nonsteroidal anti-inflammatory drugs (NSAIDs), corticosteroid injections (CSIs), and physiotherapy. Physiotherapy methods include various interventions such as manual therapy, exercise, and electrotherapy. Although these treatments do not directly treat the specific pathology, they help correct rotator cuff and scapular muscle weakness and dysfunction, reduce the tightness of the posterior capsule and other soft tissues, and relieve pain and dysfunction. It focuses on correcting the postural abnormalities that contribute to the disease.

In our study, the investigators aimed to determine the effects of rehabilitation components in the conservative treatment of patients with rotator cuff syndrome and to determine the effects of strengthening exercises on the functional status of the patients.

DETAILED DESCRIPTION:
Rotator cuff syndrome (RCS), also known as rotator cuff tendonitis, is characterised by intense pain, functional impairment, loss of shoulder range of motion (ROM), nocturnal pain, and limitations in activities of daily living. It is a common problem in the ageing population and its patophysiology may be the result of tendon degeneration resulting from microtrauma (repetitive activities, overload) or traumatic injury.

Groups Participants were randomly divided into two treatment groups. There are 10 patients in each group. The patients in the control group received a standard treatment programme, while the patients in the experimental group received strengthening exercises with theraband in addition to the standard treatment programme. Treatment sessions for both groups lasted 50-55 minutes and were performed three days a week. Details of the study groups are given below.

Control Group

Patients in the control group received a standard treatment programme. This programme included the following:

Passive stretching exercises were performed 10 repetitions for each movement (shoulder flexion, abduction, adduction, internal rotation, external rotation). Codman exercises were performed 15 repetitions (with 1kg dumbbell). Shoulder isometric exercises were performed 15 repetitions for each movement (ball press, clockwise and anti-clockwise ball rotation, finger slide on the wall). Wand exercises were performed 15 repetitions (shoulder abduction, internal rotation, external rotation). Electrotherapy was applied for 20 minutes and ice therapy was applied for 20 minutes.7-9 Experimental Group

Patients in the experimental group received strengthening exercises with theraband in addition to the standard treatment programme. This programme included the following:

Strengthening Exercises: Low-row, biceps strengthening, shoulder horizontal abduction and shoulder horizontal adduction, external rotation. After the pain decreased, strengthening exercises for subscapularis, infraspinatus, supraspinatus, teres minor, deltoid and scapulothoracic muscles were performed. The colour of the Theraband was chosen between yellow, red, green, blue and red to the extent tolerated by the patient.

ELIGIBILITY:
Inclusion Criteria:

* having complaints for at least three months
* having positive Empty can test
* having rotator cuff injury
* having loss of function in the shoulder and volunteering to participate in the study

Exclusion Criteria:

* cardiovascular disease that would interfere with the rehabilitation process,
* who had neurological or systemic musculoskeletal disease
* who had undergone upper extremity surgery
* who had upper extremity scapula fracture

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
Disability Questionnaire for Arm, Shoulder and Hand (Quick DASH): | 3 months
  Quick DASH was used as the primary outcome measure because it is a questionnaire that assesses upper extremity injuries and symptoms and measures their impact on patients' activities of daily living. Each section of the Quick-DASH questionnaire yields a score between 0 and 100 (0= no disability, 100= maximum disability).10,11

SECONDARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) | 1 months
  WORC was used to assess the impact of rotator cuff problems on quality of life.(Kirkley Alvarez) Each question is answered with a 100mm VAS. The total is between 0 and 2100, with lower scores indicating higher quality of life.
Nothingam Health Profile (NSP): | 1 months
  The NSP was used to measure the general health status and quality of life of the patients. The scoring of the sections ranges from 0-100, with higher scores indicating health problems.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin ŞAHBAZ, Study Director — Istanbul Beykent University
Locations (1):
- Physical Therapy and Rehabilitation Clinic of Istanbul Health Sciences University Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It was not considered appropriate to share individual information.

REFERENCES:
- [Background] Gomoll AH, Katz JN, Warner JJ, Millett PJ. Rotator cuff disorders: recognition and management among patients with shoulder pain. Arthritis Rheum. 2004 Dec;50(12):3751-61. doi: 10.1002/art.20668. No abstract available. PMID 15593187
- [Background] Galetta MD, Keller RE, Sabbag OD, Linderman SE, Fury MS, Medina G, O'Donnell EA, Cheng TTW, Harris E, Oh LS. Rehabilitation variability after rotator cuff repair. J Shoulder Elbow Surg. 2021 Jun;30(6):e322-e333. doi: 10.1016/j.jse.2020.11.016. Epub 2021 Jan 5. PMID 33418088